CLINICAL TRIAL: NCT04536649
Title: Proton and Heavy Ion Beam Radiation Versus Photon Beam Radiation for Newly Diagnosed Glioblastoma: A Multi-center Prospective Phase 3 Randomized Control Clinical Trial.
Brief Title: Proton and Heavy Ion Beam Radiation vs. Photon Beam Radiation for Newly Diagnosed Glioblastoma.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Collaborators: RenJi Hospital (Other); Ruijin Hospital (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Jiade J. Lu, Professor, Shanghai Proton and Heavy Ion Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-HNCNS-2020-45
Record Dates: First submitted 2020-08-25; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Carbon-ion Radiotherapy; Proton Radiotherapy; Photon Radiotherapy; Overall Survival
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard-dose Photon Radiotherapy (Experimental): The patients will receive standard-dose photon radiation (60Gy/30F for high-risk area) with concurrent temozolomide (75mg/m2, qd), adjuvant temozolomide (150-200mg/m2, qd, D1-5, 28d/cycle)
  Interventions: Radiation: Radiotherapy
- Standard-dose Proton Radiotherapy (Experimental): The patients will receive standard-dose proton radiation (60GyE/30F for high-risk area) with concurrent temozolomide (75mg/m2, qd), adjuvant temozolomide (150-200mg/m2, qd, D1-5, 28d/cycle).
  Interventions: Radiation: Radiotherapy
- Standard-dose Proton Radiotherapy plus Carbon-Ion Boost (Experimental): The patients will receive carbon-ion radiation boost (15GyE/3F for residual lesion) priot to standard-dose proton radiation (60GyE/30F for high-risk area) with concurrent temozolomide (75mg/m2, qd), then adjuvant temozolomide (150-200mg/m2, qd, D1-5, 28d/cycle).
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Multimodal brain imaging-guided radiotherapy using different beams

SUMMARY:
This is a multi-center prospective phase 3 clinical trial to explore the efficacy and side effects of standard-dose photon radiation versus standard-dose proton radiation versus carbon ion boost plus standard proton radiation for newly diagnosed glioblastoma. The patients enrolled will be randomly allocated with 1:1:1 to three group: Control Group, standard-dose photon radiotherapy; Study Group A, standard-dose proton radiotherapy; Study Group B, standard-dose proton radiotherapy plus induction carbon-ion radiotherapy boost. The primary endpoint is overall survival (OS).

DETAILED DESCRIPTION:
This multi-center prospective phase 3 clinical trial will enroll 369 patients with newly diagnosed glioblastoma. Patients will be randomly allocated with 1:1:1 to three groups: Control Group, standard-dose photon radiotherapy (60 Gy); Study Group A, standard-dose proton radiotherapy (60 GyE); Study Group B, standard-dose proton radiotherapy (60 GyE) plus induction carbon-ion radiotherapy boost (15GyE/3F). All patients will receive concurrent and adjuvant temozolomide according to the Stupp protocol. The primary endpoint is overall survival (OS). The secondary endpoint is progression-free survival, side effect and quality life.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old and <80 years old
* Pathologically confirmed newly-diagnosed GBM
* Redisual lesion after subtotal resection, partial resection, or biopsy
* No dissemination or metastasis in the spinal canal, single lesion, supratentorial lesion
* ECOG score 0-1
* Sign the informed consent form before starting the research

Exclusion Criteria:

* No pathological confirmed evidence of GBM
* Multiple lesions or distant spread indicated by imaging studies
* Receive conventional photon/proton/carbon ion radiation therapy on the head
* Received intracranial radioactive particle implantation
* A history of malignant tumors or multiple primary tumors (except skin basal cell carcinoma)
* Positive pregnancy test for women of childbearing age
* With the accompanying diseases or conditions affect the safety of patients during normal enrollment or research
* Active mental disorders or other mental disorders that affect the patients ability to sign informed consent and understand
* Uncontrolled active infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From the pathological confirmation to death, a median of 3 years.
  The interval from randomization to death

SECONDARY OUTCOMES:
Progression-free Survival | From randomization to tumor progression, with a median of 3 years.
  The interval from randomization to progression or death
Toxicities | From start to 12 months after completion of radiotherapy.
  The scores of toxicities are based on CTCAE criteria, which refers to Common Terminology Criteria for Adverse Events.
Recognitive Function | From initiation of radiotherapy to 12 months after completion of radiotherapy.
  The assessment of recognitive function is based on MMSE criteria, which refers to Mini-Mental State Examination.
Life Quality | From initiation of radiotherapy to 12 months after completion of radiotherapy.
  The assessment of life quality is based on ADL criteria, which refers to Activities of Daily Living.

CONTACTS AND LOCATIONS:
Overall Officials: Jiade J Lu, Principal Investigator — Shanghai Proton and Heavy Ion Center
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data will be uploaded by excel documents to share the IPD.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: On March, 2026
Access Criteria: Excel document as the repository will be used for management.